CLINICAL TRIAL: NCT05767151
Title: The Chinese DENOVO Parkinson's Disease Registry
Brief Title: Chinese DENOVO PD Registry
Status: Recruiting | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: CPD-DENOVOR
Record Dates: First submitted 2022-08-29; First posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2022-08

CONDITIONS: Parkinson Disease
Keywords: Motor symptoms; Nonmotor symptoms; Chinese longitudinal cohort; disease progression; biomarker
MeSH Terms: conditions — Parkinson Disease; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Extraction of DNA from peripheral blood of patients
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of this longitudinal, multi-center study is to explore the clinical characteristics of PD and confirm biomarkers for PD evolution or progression.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a common neurodegenerative disease, characterized by classical motor features including tremor, rigidity, bradykinesia, postural instability and a wide range of non-motor symptoms. Notably, a good deal of research revealed that PD is heterogeneous in clinical manifestations, rate of progression and prognosis. It is crucial to acknowledge the marked heterogeneity of PD and establish compelling biomarkers to predict the disease progression and prognosis. In past decades, there were substantial studies focused on defining the biomarkers of PD, which substantially contributed to improving our knowledge of PD. However, the pathology and clinical heterogeneity of PD are still poorly understood and controversial. Moreover, the information about reliable and well-validated biomarkers for PD has not yet been investigated thoroughly. Investigators aim to characterize the clinical feature, genetic basis, environmental factors and their interactions among different PD subtypes in China, and identify promising biomarkers for PD progression.

Data were collected at baseline, 12±1 months during the routine follow-up visits. Information about detailed disease history, level of education, significant chronic comorbidities, physical examination, medication history, family history, living habits and toxic exposure history, which include smoking, drinking tea, alcoholic consumption, drinking coffee, exposure to pesticide or occupational solvent, history of carbon monoxide poisoning and recurrent head trauma will be recorded at baseline. For each visit evaluation, the same questionnaires will be conducted. A standardized neurological assessment according to the recommendation of Consensus on the construction of clinical database of Parkinson's disease and movement disorders in China. The Unified Parkinson's Disease Rating Scale (UPDRS) part III is conducted for motor assessment, all the patients are evaluated in "OFF" state. The clinical stage of PD is assessed by Hoehn and Yahr scale (H-Y). The non-motor symptoms are evaluated by Non-motor Symptom Scale (NMSS), autonomic symptoms are evaluated by The Scale for outcomes in Parkinson's disease for Autonomic Symptoms (SCOPA-AUT). Constipation was diagnosed by Functional Constipation Diagnostic Criteria Rome. The 39-item Parkinson's Disease Questionnaire (PDQ-39) was used to assess the quality of life. Sleep quality was evaluated by Parkinson's Disease Sleep Scale (PDSS) and excessive daytime sleepiness by Epworth Sleepiness Scale (ESS). Probable rapid eye movement sleep behavior disorder (p-RBD) was diagnosed by rapid eye movement sleep behavior questionnaire-Hongkong (RBDQ-HK). Restless leg syndrome (RLS) was diagnosed with the Cambridge Hopkins Restless Leg syndrome questionnaire (CH-RLSq). Cognition was used by the previously validated scale, Mini Mental State Examination (MMSE) and Montreal Cognitive Assessment (MoCA). Olfaction test was carried out by Hyposmia Rating Scale (HRS), and a proportion of patients was also ascertained by Sniffin's Sticks. Depression was diagnosed by Hamilton Depression Scale (HAMD). Symptom of fatigue was measured by PD fatigue severity scale (PFS). Wearing-off was evaluated by WOQ-9 and freezing gait by new freezing gait questionnaire scores (NFOGQ). Dyskinesis was evaluated by Rush Dyskinesia Rating Scale. DNA samples were extracted from peripheral blood and detected by Whole Exome Sequencing or Whole-genome sequencing. Plasma was obtained from venepuncture. All the participants were scanned by structural MRI to exclude obvious intracranial lesions and other parkinsonism such as MSA, PSP and WD.

ELIGIBILITY:
Inclusion Criteria:

1. Participants were diagnosed by MDS Clinical Diagnostic Criteria for PD
2. Disease duration ≤ 2 years at baseline
3. Hoehn-Yahr stage ≤2 at baseline
4. The age of PD patients ranges from 30 to 75 years old
5. Participants were naive to antiparkinsonian therapy
6. Able to Written informed consent

Exclusion Criteria:

1. Participants were diagnosed with parkinsonism-syndrome
2. Participants were treated with antiparkinsonian drugs at baseline
3. Participants with cognitive impairment
4. Unable to Written informed consent

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study Population: Most of the PD patients come from mainland China, especially from Hunan Province, Hubei Province, Jiangxi Province and Guizhou Province. The age of PD patients ranges from 30 to 75 years old.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2031-01-01 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
The Unified Parkinson's Disease Rating Scale for evaluating motor subtypes | from baseline to 10 years
  The UPDRS is made up of four parts, 55 items in total. Total score varies from 0 to 199. Part I: evaluation of behavior and mood, which consists of 4 items, score varies from 0-16; Part II: self-evaluation of the activities of daily life, which consists of 13 items,score varies from 0-52; Part III: motor evaluation, which consists of 27 items, score varies from 0-108; Part IV: complications of therapy, which consists of 11 items,score varies from 0-23. All the patients are evaluated in "OFF" state. The ratio of the mean tremor score (scores of item-16, item-20, and item-21 will be added: ) to the mean postural instability/gait disorder (PIGD) score (scores of item-13, item-14, item-15, item-29, item-30 will be added: ) was used to classify motor subtype. Patients with a ratio value < 1.0 were defined as PIGD, and those with values from 1.0 to 1.5 were categorized as intermediate, while those with values ≥1.5 were classified as tremor dominant.
The clinical stage of PD is assessed by Hoehn and Yahr scale | from baseline to 10 years
  The H-Y scale ranges from 1 to 5. Early PD is defined as H-Y stage 1 to 2.5, advanced PD is defined as H-Y stage 3-5.
The non-motor symptoms are evaluated by Non-motor Symptom Scale | from baseline to 10 years
  This scale includes 30 items which is divided into 9 domains. Total score varies from 0-360. Higher score indicates severer symptoms. Domain 1 evaluates cardiovascular system symptoms. Score of domain 1 varies from 0-24.
  Domain 2 evaluates sleep condition. Score of domain 2 varies from 0-48. Domain 3 evaluates cognitive function. Score of domain 3 varies from 0-72. Domain 4 evaluates illusion. Score of domain 4 varies from 0-36. Domain 5 evaluates attention and memory. Score of domain 5 varies from 0-36. Domain 6 evaluates gastrointestinal symptoms. Score of domain 6 varies from 0-36. Domain 7 evaluates urinary symptoms. Score of domain 7 varies from 0-36. Domain 8 evaluate sensory symptoms. Score of domain 8 varies from 0-24. Domain 9 evaluates other non-motor symptoms.
  Score of domain 9 varies from 0-48.
Constipation was diagnosed by Functional Constipation Diagnostic Criteria Rome III | from baseline to 10 years
  The diagnostic criteria must include two or more of the following
  1. Straining during at least 25% of defecations
  2. Lumpy or hard stools in at least 25% of defecations
  3. Sensation of incomplete evacuation for at least 25% of defecations
  4. Sensation of anorectal obstruction/blockage for at least 25% of defecations
  5. Manual maneuvers to facilitate at least 25% of defecations (e.g., digital evacuation, support of the pelvic floor)f. Fewer than three defecations per week 2. Loose stools are rarely present without the use of laxatives 3.
  Insufficient criteria for irritable bowel syndrome * Criteria fulfilled for the last 3 months with symptom onset at least 6 months prior to diagnosis
The PDQ-39 was used to assess the quality of life | from baseline to 10 years
  This scale includes 39 items assessing the following regions: mobility (10 items), activities of daily living (6 items), emotional well-being (6 items), stigma (4 items), social support (3 items), cognitions (4 items), communications (3 items) and bodily discomfort (3 items). Alternatively, the sum of the scores can assess the overall health-related quality of life profile of the individual questioned. Scores in each region should be added. The score of the answers ranges from 0 to 4 for each item and the total score ranges from 0 to 116, where higher scores reflect worse life quality
Sleep quality is evaluated by Parkinson's Disease Sleep Scale | from baseline to 10 years
  This scale includes 15 items that address eight aspects of sleep disturbances in PD, including overall quality of night's sleep (item 1)), score of item 1 less than 6 is defined as sleep disorder. Score of all the questions will be summed. The score of the answers ranges from 0 to 10 for each item and the total score ranges from 0 to 150, where higher scores reflect better sleep condition.
Epworth Sleepiness Scale evaluates excessive sleepiness | from baseline to 10 years
  This scale includes 8 items. Score of all the questions will be summed. All items were rated on a 4-point scale (0- 3), with a minimal score of 0, and maximum total score of 24. A higher score demonstrates more severe excessive daytime sleepiness. Participants were classified as showing excessive daytime sleepiness if their total score ≥10 .
Probable rapid eye movement sleep behavior disorder was diagnosed by Probable rapid eye movement sleep behavior disorder Questionnaire -Hongkong | from baseline to 10 years
  This scale includes 13 items. Score of all the questions will be summed. Total score of the answers ranges from 0 to 100, where higher scores reflect severer rapid eye movement sleep behavior disorder.The optimal cutoff value for the overall scale is 17; subjects were classified as showing RBD when they reached the above score.
Olfaction test was measured by Hyposmia Rating Scale | from baseline to 10 years
  This scale includes 6 items. Score of all the questions will be summed. All items were rated on a 4-point scale (1-4), with a minimal score of 6, and maximum total score of 24. A higher score demonstrates more worse sense of olfaction.
  The cutoff value HRS is 22.5.
Cognitive condition is assessed by Mini Mental State Examination | from baseline to 10 years
  This scale includes 30 items. Score of all the questions will be summed. All items were rated on a 2-point scale (0-
  1), with a minimal score of 0, and maximum total score of 30. A higher score demonstrates more better cognitive condition. The definition of cognitive disorder differs in education level. For illiteracy, presence of cognitive impairment is defined as MMSE score. For those only receive elementary education, the cut-off value is 20. For other patients, presence of cognitive impairment was defined as MMSE scores less than 25.
Depression was diagnosed by Hamilton and Montgomery-Asberg Depression Scale | from baseline to 10 years
  This scale includes 17 items. Score of all the questions will be summed. Total score ranges from0-53. A higher score demonstrates more severer depression. The study participants were defined to be not depressed (scores 0-6) , to have minor depression(scores 7-14), or to have major depression (scores above 14) at the different visits during follow-up.
Autonomic symptoms are evaluated by The Scale for outcomes in Parkinson disease for Autonomic Symptoms | from baseline to 10 years
  This scale includes 25 items assessing the following regions: gastrointestinal (7 items), urinary (6 items), cardiovascular (3 items), thermoregulatory (4 items), pupillomotor (1 items), and sexual dysfunction(2 items for men and 2 items for women). Scores in each region should be added. The score of the answers ranges from 0 to 3 for each item and the total score ranges from 0 to 69, where higher scores reflect worse autonomic functioning.
Restless leg syndrome (RLS) was diagnosed with the Cambridge Hopkins Restless Leg syndrome questionnaire | from baseline to 10 years
  1. have, or have you had, recurrent uncomfortable feelings or sensations in your legs while you are sitting or lying down
  2. have, or have you had, a recurrent need or urge to move your legs while you were sitting or lying down
  3. more likely to have these feelings when you are resting
  4. If you get up or move around when you have these feelings, these feelings get better
  5. these feelings in your legs most likely to occur at mid-day or afternoon or evening or night
  6. Simply changing leg position by itself once without continuing to move usually relieve these feelings usually don't relieves
  7. These feelings are not or not always due to muscle cramps
Symptom of fatigue was measured by PD fatigue severity scale | from baseline to 10 years
  This scale includes 9 items. Score of all the questions will be summed. All items were rated on a 7-point scale (1-7).
  Total score ranges from0-63. A higher score demonstrates more severer fatigue.
Freezing gait by new freezing gait questionnaire scores | from baseline to 10 years
  Parts II and III provides a total summed score between 0 and 28. Part II (items 2-6, scoring range 0-19) rated the severity of FOG based on its duration and frequency in its most common manifestation. Total score will be calculated for comparison.
Dyskinesia was evaluated by UPDRS part III | from baseline to 10 years
  The presence of dyskinesia is evaluated by the doctor and recordsed.

SECONDARY OUTCOMES:
Comparison between Rates of Change | from baseline to 10 years
  Comparison between the rates of change in the mean of clinical outcomes in PD subtype, inluding postural instability/gait disorder (PIGD), intermediate, and tremor dominant (TD).

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital of Central South University, Changsha, Hunan, China